CLINICAL TRIAL: NCT00488475
Title: A 1 Year Observational Study of the Use of Etanercept in Routine German Clinical Practice to Treat Rheumatoid Arthritis Patients: a Health Economic, Safety and Effectiveness Evaluation
Brief Title: Observational Trial With Enbrel
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A1-102335; B1801121
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Rheumatoid Arthritis
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — The patients will be treated in accordance with the requirements of the labelling of Enbrel® in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.
  Other Names: Enbrel

SUMMARY:
The diagnosis, evaluation and treatment of rheumatoid arthritis (RA) continue to undergo rapid change. Randomized controlled trials such as the TEMPO study have demonstrated the efficacy and safety of the combination of etanercept and methotrexate. Importantly, the TEMPO study showed that patients treated with etanercept and methotrexate could reach the newer therapeutic goals of low disease activity and remission, and that the physicians, patients, and payers are no longer prepared to accept the goal of "Reduction of symptoms". RCT are important and powerful tools in assessing efficacy and safety but have their limitations in terms of generalisability. In order to assess health economics, clinical effectiveness and safety of etanercept, they need to be measured by performing observational studies of unselected patients. This study aims to provide a holistic assessment of patients receiving etanercept in a real world setting. This will include centers that would not normally take part in RCT. The study will assess treatment with etanercept with descriptive statistics of the following parameters: Health economic, Safety, Effectiveness. In addition, there was a previous study of similar design, but of only 3 months duration (101354), which will allow comparison with historical data. Since previous study, there have been a number of significant changes: Introduction of a new formulation for etanercept (Enbrel® 50mg · once weekly), Definition of early RA has been modified to short disease duration (from 3 months to 1 year).

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rheumatoid arthritis

Exclusion Criteria:

* Sepsis or risk for sepsis,
* Acute infection,
* Hypersensitivity against Etanercept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients for whom the decision has already been made to initiate treatment with Enbrel® can be enrolled in this observational trial. These patients must have a proven diagnosis of Rheumatoid Arthritis
Sampling Method: Non-Probability Sample
Enrollment: 4945 (Actual)
Dates: Start 2006-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Druce KL, Aikman L, Dilleen M, Burden A, Szczypa P, Basu N. Fatigue independently predicts different work disability dimensions in etanercept-treated rheumatoid arthritis and ankylosing spondylitis patients. Arthritis Res Ther. 2018 May 29;20(1):96. doi: 10.1186/s13075-018-1598-8. PMID 29843776
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-102335&StudyName=Observational%20Trial%20with%20Enbrel

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants greater than or equal to (>=) 18 years of age, who had confirmed diagnosis of moderate to severe rheumatoid arthritis (RA) and received etanercept (Enbrel) as per German Summary of Product Characteristics (SPC), were observed prospectively up to Week 52.
Period: Overall Study
Arm/Group | Etanercept
Started | 4945
Completed | 3191
Not Completed | 1754
Not completed — Other | 1754

BASELINE CHARACTERISTICS:
Population: Safety population included all participants with available documentations.
Arm/Group | Etanercept
Number analyzed (Participants) | 4871
Age, Continuous [Mean (Standard Deviation); unit: years] — Evaluable participants for this Baseline measure were 4868.
  years | 55.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3652
  Male | 1219

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Functional Remission Determined by Hannover Functional Ability Questionnaire (FFbH) at Week 26
Description: Hannover Functional Ability Questionnaire (FFbH) consists 18 questions to assess daily activities in last 7 days. Each question is answered by the participant as "Yes, I can perform the activity without difficulty" (score assigned = 2), "Yes, but with some difficulties" (score assigned = 1) and "No or only with help" (score assigned = 0). Final FFbH score (FFbH functional capacity) is then computed according to formula: (Sum of all single scores * 100% [percent]) / (2 * number of answered questions) ranging between 0-100; higher score indicates better daily activities. FFbH functional remission is defined as FFbH functional capacity of >= 83%.
Time Frame: Week 26
Population: Effectiveness population included all participants >= 18 years of age, confirmed diagnosis of rheumatoid arthritis, who had not received treatment with etanercept previously and who had post baseline documentations. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 3723
percentage of participants | 36.4 [34.8 to 37.9]

2. Primary Outcome: Percentage of Participants Achieving Functional Remission Determined by Hannover Functional Ability Questionnaire (FFbH) at Week 52
Description: Hannover Functional Ability Questionnaire (FFbH) consists 18 questions to assess daily activities in last 7 days. Each question is answered by the participant as "Yes, I can perform the activity without difficulty" (score assigned = 2), "Yes, but with some difficulties" (score assigned = 1) and "No or only with help" (score assigned = 0). Final FFbH score (FFbH functional capacity) is then computed according to formula: (Sum of all single scores * 100%) / (2 * number of answered questions), ranging between 0-100; higher score indicates better daily activities. FFbH functional remission is defined as FFbH functional capacity of >= 83%.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 3085
percentage of participants | 41.5 [39.7 to 43.2]

3. Secondary Outcome: Euro Quality of Life-5 Dimensions (EQ-5D) Visual Analog Scale (VAS)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 millimeter (mm) (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Week 26, Week 52
Population: Effectiveness population included all participants >= 18 years of age, confirmed diagnosis of RA, who had not received treatment with etanercept previously and who had post baseline documentations. Here 'N' (number of participants analyzed) = participants evaluable for this measure and 'n' = participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 4718
mm
  Baseline (n = 4718) | 53.1 (21.3)
  Week 26 (n = 3637) | 66.5 (20.7)
  Week 52 (n = 3036) | 70.0 (20.5)

4. Secondary Outcome: Euro Quality of Life-5 Dimensions (EQ-5D) Time Trade Off (TTO)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health state profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain or discomfort, and anxiety or depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQol group assigns a utility value for each domain in the profile. EQ-5D score is transformed to EQ-5D-TTO score ranging from -0.205 to 0.999; higher score indicates a better health state.
Time Frame: Baseline, Week 26, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 4718
units on a scale
  Baseline (n = 4718) | 0.579 (0.302)
  Week 26 (n = 3637) | 0.748 (0.244)
  Week 52 (n = 3036) | 0.782 (0.227)

5. Secondary Outcome: Work Productivity and Activity Impairment - Special Health Problems (WPAI:SHP)
Description: WPAI:SHP is 6-question participant rated questionnaire to determine the amount of absenteeism, presenteeism, work productivity loss and daily activity impairment attributable to rheumatoid arthritis for a period of 7 days prior to each visit. It yields 4 sub-scores: work time missed (absenteeism), impairment while working (presenteeism or reduced on-the-job effectiveness), overall work impairment (work productivity loss or absenteeism plus presenteeism) and activity impairment (daily activity impairment). These sub-scores are transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Baseline, Week 26, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Etanercept
Number analyzed (Participants) | 4716
percentage of impairment
  Baseline: Work Time Missed (n = 1295) | 22.5 (37.0)
  Baseline: Impairment While Working (n = 1534) | 49.5 (27.1)
  Baseline: Overall work impairment (n = 1173) | 54.1 (29.0)
  Baseline: Activity impairment (n = 4716) | 60.7 (23.2)
  Week 26: Work Time Missed (n = 946) | 9.4 (25.8)
  Week 26: Impairment While Working (n = 1267) | 31.1 (24.5)
  Week 26: Overall work impairment (n = 909) | 33.0 (26.9)
  Week 26: Activity impairment (n = 3640) | 42.0 (24.7)
  Week 52: Work Time Missed (n = 815) | 9.1 (25.1)
  Week 52: Impairment While Working (n = 1076) | 27.8 (23.2)
  Week 52: Overall work impairment (n = 790) | 30.9 (26.1)
  Week 52: Activity impairment (n = 3011) | 38.0 (24.1)

6. Secondary Outcome: Healthcare Resource Utilization
Description: Participants' utilization of healthcare resources was evaluated as number of events for healthcare resources utilization including: number of visits to general practitioners, visits to rheumatologist, visits to other medical specialists, inpatient hospitalizations, inpatient rehabilitations, inpatient follow-up treatment, outpatient rehabilitations, physiotherapy, and other healthcare utilizations. At baseline, number of events for participants' healthcare resources utilization during last 12 months before enrollment into the study were documented. After enrollment, number of events for participants' healthcare resources utilization were documented for last 6 months after previous documentation.
Time Frame: Baseline, Week 26, Week 52
Population: Effectiveness population. Here 'N' (number of participants analyzed) = overall participants evaluable for any event for this measure and 'n'= participants evaluable for specified event at specified time points.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Etanercept
Number analyzed (Participants) | 4727
events
  Baseline: General Practitioner Visit (n = 4034) | 7.4 (8.2)
  Baseline: Rheumatologist Visit (n = 4345) | 6.0 (5.0)
  Baseline: Other Specialist Visit (n = 3034) | 3.1 (5.4)
  Baseline: In-patient Hospitalization (n = 2622) | 0.9 (2.7)
  Baseline: In-patient Rehabilitation (n = 2047) | 0.4 (2.6)
  Baseline: Follow-up Treatment (n = 1861) | 0.1 (1.7)
  Baseline: Out-patient Rehabilitation (n = 1854) | 0.1 (1.3)
  Baseline: Physiotherapy (n = 2577) | 9.8 (21.5)
  Baseline: Other Health Care Resources (n = 1169) | 3.0 (13.5)
  Week 26: General Practitioner Visit (n = 3139) | 3.6 (4.4)
  Week 26: Rheumatologist Visit (n = 3424) | 3.8 (3.2)
  Week 26: Other Specialist Visit (n = 2432) | 1.3 (1.9)
  Week 26: In-patient Hospitalization (n = 1893) | 0.2 (1.0)
  Week 26: In-patient Rehabilitation (n = 1772) | 0.2 (1.5)
  Week 26: Follow-up Treatment (n = 1692) | 0.0 (0.6)
  Week 26: Out-patient Rehabilitation (n = 1675) | 0.1 (1.5)
  Week 26: Physiotherapy (n = 2095) | 4.9 (11.8)
  Week 26: Other Health Care Resources (n = 1251) | 1.5 (9.7)
  Week 52: General Practitioner Visit (n = 2622) | 3.0 (3.8)
  Week 52: Rheumatologist Visit (n = 2859) | 2.6 (2.3)
  Week 52: Other Specialist Visit (n = 2013) | 1.3 (1.8)
  Week 52: In-patient Hospitalization (n = 1583) | 0.2 (0.9)
  Week 52: In-patient Rehabilitation (n = 1485) | 0.1 (1.4)
  Week 52: Follow-up Treatment (n = 1451) | 0.0 (1.1)
  Week 52: Out-patient Rehabilitation (n = 1440) | 0.0 (0.5)
  Week 52: Physiotherapy (n = 1746) | 4.8 (11.3)
  Week 52: Other Health Care Resources (n = 1064) | 1.1 (6.3)

7. Secondary Outcome: Duration of Healthcare Resources Utilization
Description: Participants' duration of healthcare resources utilization was evaluated as number of days for healthcare resources utilization including: duration of visits to general practitioners, to rheumatologist, to other medical specialists, inpatient hospitalizations, inpatient rehabilitations, inpatient follow-up treatment, outpatient rehabilitations, physiotherapy, and other healthcare utilizations. At baseline, number of days for participants' healthcare resources utilizations during last 12 months before enrollment into the study were documented. After enrollment, number of days for participants' healthcare resources utilization were documented for last 6 months after previous documentation.
Time Frame: Baseline, Week 26, Week 52
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Etanercept
Number analyzed (Participants) | 2989
days
  Baseline: General Practitioner Visit (n = 1752) | 4.0 [0.0 to 104.0]
  Baseline: Rheumatologist Visit (n = 1916) | 4.0 [0.0 to 50.0]
  Baseline: Other Specialist Visit (n = 1381) | 2.0 [0.0 to 150.0]
  Baseline: In-patient Hospitalization (n = 1747) | 7.0 [0.0 to 160.0]
  Baseline: In-patient Rehabilitation (n = 1030) | 0.0 [0.0 to 60.0]
  Baseline: Follow-up Treatment (n = 826) | 0.0 [0.0 to 49.0]
  Baseline: Out-patient Rehabilitation (n = 838) | 0.0 [0.0 to 65.0]
  Baseline: Physiotherapy (n = 1333) | 6.0 [0.0 to 365.0]
  Baseline: Other Health Care Resources (n = 645) | 0.0 [0.0 to 156.0]
  Week 26: General Practitioner Visit (n = 1505) | 2.0 [0.0 to 50.0]
  Week 26: Rheumatologist Visit (n = 1649) | 3.0 [0.0 to 48.0]
  Week 26: Other Specialist Visit (n = 1201) | 0.0 [0.0 to 20.0]
  Week 26: In-patient Hospitalization (n = 1113) | 0.0 [0.0 to 90.0]
  Week 26: In-patient Rehabilitation (n = 977) | 0.0 [0.0 to 38.0]
  Week 26: Follow-up Treatment (n = 893) | 0.0 [0.0 to 28.0]
  Week 26: Out-patient Rehabilitation (n = 883) | 0.0 [0.0 to 90.0]
  Week 26: Physiotherapy (n = 1211) | 0.0 [0.0 to 104.0]
  Week 26: Other Health Care Resources (n = 817) | 0.0 [0.0 to 180.0]
  Week 52: General Practitioner Visit (n = 1255) | 2.0 [0.0 to 52.0]
  Week 52: Rheumatologist Visit (n = 1379) | 2.0 [0.0 to 21.0]
  Week 52: Other Specialist Visit (n = 999) | 0.0 [0.0 to 16.0]
  Week 52: In-patient Hospitalization (n = 947) | 0.0 [0.0 to 112.0]
  Week 52: In-patient Rehabilitation (n = 829) | 0.0 [0.0 to 50.0]
  Week 52: Follow-up Treatment (n = 791) | 0.0 [0.0 to 37.0]
  Week 52: Out-patient Rehabilitation (n = 789) | 0.0 [0.0 to 90.0]
  Week 52: Physiotherapy (n = 1022) | 0.0 [0.0 to 104.0]
  Week 52: Other Health Care Resources (n = 698) | 0.0 [0.0 to 90.0]

8. Secondary Outcome: Duration of Working Disability
Description: Duration of working disability was assessed as number of days a participant was disable to work. Duration of work disability was considered as "0" if participant was not disable to work during period of assessment. At baseline, participants' duration of working disability during last 12 months before enrollment into the study was documented. After enrollment, participants' duration of working disability was documented for last 6 months after previous documentation.
Time Frame: Baseline, Week 26, Week 52
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Etanercept
Number analyzed (Participants) | 3928
days
  Baseline (n = 3928) | 0.0 [0.0 to 365.0]
  Week 26 (n = 3168) | 0.0 [0.0 to 200.0]
  Week 52 (n = 2651) | 0.0 [0.0 to 200.0]

9. Secondary Outcome: Disease Activity Score Based on 28-Joints Count (DAS28)
Description: DAS28 calculated from the number of swollen joints (SJC) and tender joints (TJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and Patient global assessment of disease activity (recorded on a VAS of 0 mm [very good] to 100 mm [very bad]). Total score range: 0 to 10, higher score indicated more disease activity. DAS28 less than (<) 2.6 = remission, DAS28 less than or equal to (<=) 3.2 = low disease activity, DAS28 greater than or equal to (>=) 3.2 to <=5.1 = moderate disease activity, DAS28 greater than (>) 5.1 = high disease activity.
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 4304
units on a scale
  Baseline (n = 4304) | 5.4 (1.3)
  Week 2 (n = 2558) | 4.2 (1.5)
  Week 6 (n = 3212) | 3.9 (1.5)
  Week 12 (n = 3363) | 3.7 (1.5)
  Week 26 (n = 3116) | 3.6 (1.5)
  Week 38 (n = 2719) | 3.4 (1.4)
  Week 52 (n = 2608) | 3.3 (1.4)

10. Secondary Outcome: Swollen Joints Count (SJC)
Description: Number of swollen joints was determined by examination of 28 joints and identifying when swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Etanercept
Number analyzed (Participants) | 4804
joints
  Baseline (n = 4804) | 7.0 (5.8)
  Week 2 (n = 4091) | 4.5 (5.1)
  Week 6 (n = 4251) | 3.4 (4.4)
  Week 12 (n = 4209) | 3.0 (4.2)
  Week 26 (n = 3764) | 2.6 (3.9)
  Week 38 (n = 3302) | 2.4 (3.7)
  Week 52 (n = 3110) | 2.0 (3.3)

11. Secondary Outcome: Tender Joints Count (TJC)
Description: Number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Etanercept
Number analyzed (Participants) | 4820
joints
  Baseline (n = 4820) | 9.7 (7.3)
  Week 2 (n = 4099) | 6.5 (6.7)
  Week 6 (n = 4259) | 5.0 (5.9)
  Week 12 (n = 4216) | 4.4 (5.8)
  Week 26 (n = 3790) | 3.9 (5.4)
  Week 38 (n = 3313) | 3.5 (5.2)
  Week 52 (n = 3129) | 3.1 (4.8)

12. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. Normal range is 0-30 mm/hour. A higher rate is consistent with inflammation.
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter per hour (mm/h)
Arm/Group | Etanercept
Number analyzed (Participants) | 4358
millimeter per hour (mm/h)
  Baseline (n = 4358) | 32.3 (23.3)
  Week 2 (n = 2634) | 24.4 (20.0)
  Week 6 (n = 3297) | 24.0 (19.6)
  Week 12 (n = 3456) | 24.0 (20.2)
  Week 26 (n = 3198) | 23.6 (19.7)
  Week 38 (n = 2782) | 23.1 (19.9)
  Week 52 (n = 2665) | 22.4 (18.9)

13. Secondary Outcome: Percentage of Participants With Remission Determined by Disease Activity Score Based on 28-Joints Count (DAS 28)
Description: DAS28 calculated from the number of swollen joints (SJC) and tender joints (TJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and Patient global assessment of disease activity (recorded on a VAS of 0 mm [very good] to 100 mm [very bad]). Total score range: 0 to 10, higher score indicated more disease activity. DAS28 defined remission was classified as a score of <2.6.
Time Frame: Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 3363
percentage of participants
  Week 2 (n = 2558) | 15.1 [13.7 to 16.5]
  Week 6 (n = 3212) | 20.8 [19.4 to 22.2]
  Week 12 (n = 3363) | 24.9 [23.5 to 26.4]
  Week 26 (n = 3116) | 28.3 [26.7 to 29.9]
  Week 38 (n = 2719) | 32.3 [30.5 to 34.0]
  Week 52 (n = 2608) | 35.2 [33.3 to 37.0]

14. Secondary Outcome: Percentage of Participants With Response Determined by Disease Activity Score Based on 28-Joints Count (DAS 28)
Description: The DAS28-based European League Against Rheumatism (EULAR) response criteria was used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and level of disease activity reached (final values). Good responders: change from baseline >1.2 with DAS28 final value <=3.2; moderate responders: change from baseline >1.2 with DAS28 final values >3.2 to <=5.1 and >5.1 or change from baseline >0.6 to <=1.2 with DAS28 final values <=3.2 and >3.2 to <=5.1; non-responders: change from baseline <=0.6 with DAS28 final values <=3.2, >3.2 to <=5.1 and >5.1 or change from baseline >0.6 to <=1.2 with DAS28 final values >5.1. Good and moderate responders were considered to have DAS28 response.
Time Frame: Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 3097
percentage of participants
  Week 2 (n = 2366) | 60.7 [58.7 to 62.7]
  Week 6 (n = 2967) | 69.7 [68.0 to 71.4]
  Week 12 (n = 3097) | 72.9 [71.3 to 74.5]
  Week 26 (n = 2866) | 77.1 [75.5 to 78.6]
  Week 38 (n = 2513) | 78.2 [76.6 to 79.8]
  Week 52 (n = 2415) | 81.7 [80.1 to 83.2]

15. Secondary Outcome: Duration of Morning Stiffness
Description: Duration of morning stiffness was defined as the time elapsed when participant woke up in the morning and was able to resume normal activities without stiffness in minutes (If none was present = 0; If stiffness persisted the entire day, 999 minutes was recorded [largest value possible to document] which may also include values up to 1440 minutes [= complete day]).
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Median (Full Range); unit: minutes
Arm/Group | Etanercept
Number analyzed (Participants) | 4763
minutes
  Baseline (n = 4763) | 60.0 [0.0 to 999.0]
  Week 2 (n = 4168) | 30.0 [0.0 to 999.0]
  Week 6 (n = 4293) | 20.0 [0.0 to 999.0]
  Week 12 (n = 4228) | 15.0 [0.0 to 999.0]
  Week 26 (n = 3792) | 15.0 [0.0 to 999.0]
  Week 38 (n = 3315) | 10.0 [0.0 to 999.0]
  Week 52 (n = 3131) | 10.0 [0.0 to 720.0]

16. Secondary Outcome: Patient Global Assessment of Arthritis Pain
Description: Participants assessed arthritis pain using a 0 mm - 100 mm Visual Analog Scale (VAS) where 0 mm = minimum possible pain (best) and 100 mm = maximum possible pain (worst).
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 4828
mm
  Baseline (n = 4828) | 64.6 (20.7)
  Week 2 (n = 4194) | 45.2 (24.0)
  Week 6 (n = 4321) | 39.2 (24.4)
  Week 12 (n = 4263) | 36.9 (25.0)
  Week 26 (n = 3818) | 35.3 (24.4)
  Week 38 (n = 3352) | 33.2 (24.4)
  Week 52 (n = 3150) | 30.8 (23.4)

17. Secondary Outcome: Physician Global Assessment of Disease Activity
Description: Physician global assessment of disease activity was measured on a 0 mm to 100 mm Visual Analog Scale (VAS), with 0 mm = no disease activity and 100mm = maximum possible disease activity.
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 4800
mm
  Baseline (n = 4800) | 61.7 (17.7)
  Week 2 (n = 4151) | 43.6 (21.4)
  Week 6 (n = 4279) | 35.6 (21.2)
  Week 12 (n = 4224) | 31.8 (21.3)
  Week 26 (n = 3787) | 30.1 (20.7)
  Week 38 (n = 3322) | 27.1 (20.4)
  Week 52 (n = 3125) | 24.7 (19.2)

18. Secondary Outcome: Patient Global Assessment of Disease Activity
Description: Patient global assessment of disease activity was measured using a 100 mm Visual Analog Scale (VAS) ranging from 0 mm= very good to 100 mm = very bad.
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 4835
mm
  Baseline (n = 4835) | 64.0 (19.7)
  Week 2 (n = 4197) | 46.6 (22.5)
  Week 6 (n = 4325) | 39.9 (23.1)
  Week 12 (n = 4268) | 37.0 (23.6)
  Week 26 (n = 3823) | 34.9 (23.2)
  Week 38 (n = 3351) | 32.6 (23.3)
  Week 52 (n = 3158) | 30.2 (22.3)

19. Secondary Outcome: C-Reactive Protein (CRP)
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 2, 6, 12, 26, 38, 52
Population: Safety analysis population included all participants with available documentations. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Etanercept
Number analyzed (Participants) | 4301
milligram per deciliter (mg/dL)
  Baseline (n = 4301) | 2.1 (2.8)
  Week 2 (n = 2524) | 1.2 (2.2)
  Week 6 (n = 3204) | 1.3 (2.3)
  Week 12 (n = 3422) | 1.2 (2.2)
  Week 26 (n = 3166) | 1.2 (2.2)
  Week 38 (n = 2773) | 1.2 (2.1)
  Week 52 (n = 2650) | 1.1 (1.9)

20. Secondary Outcome: Fatigue Visual Analog Scale (VAS)
Description: Participants assessed their fatigue during the last 7 days using a 0 mm - 100 mm VAS, where 0 mm = no fatigue and 100 mm = worst possible fatigue.
Time Frame: Baseline, Week 26, 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept
Number analyzed (Participants) | 4818
mm
  Baseline (n = 4818) | 59.8 (24.4)
  Week 26 (n = 3797) | 36.0 (26.2)
  Week 52 (n = 3140) | 32.3 (25.9)

21. Other Pre Specified Outcome: Percentage of Participants With Low Disease Activity Determined by Disease Activity Score 28 Based on 28-joints Count (DAS 28)
Description: DAS28 calculated from the number of swollen joints (SJC) and tender joints (TJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and Patient global assessment of disease activity (recorded on a VAS of 0 mm [very good] to 100 mm [very bad]). Total score range: 0 to 10, higher score indicated more disease activity. DAS28 defined low disease activity was classified as a score of <=3.2.
Time Frame: Week 2, 6, 12, 26, 38, 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 3363
percentage of participants
  Week 2 (n = 2558) | 28.0 [26.3 to 29.8]
  Week 6 (n = 3212) | 35.4 [33.8 to 37.1]
  Week 12 (n = 3363) | 40.3 [38.6 to 41.9]
  Week 26 (n = 3116) | 44.1 [42.3 to 45.9]
  Week 38 (n = 2719) | 47.4 [45.5 to 49.3]
  Week 52 (n = 2608) | 51.5 [49.6 to 53.4]

22. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included SAEs as well as non-serious AEs which occurred during the study.
Time Frame: Week 2 up to Week 52
Population: Safety analysis population included all participants with available documentations.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 4871
participants
  AEs | 2259
  SAEs | 649

23. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) With or Without Concomitant Methotrexate (MTX) Therapy
Description: Participants with or without concomitant methotrexate (MTX) treatment were reported for AEs or SAEs. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Week 2 up to Week 52
Population: Safety analysis population included all participants with available documentations. Here 'N' (number of participants analyzed) signifies participants evaluable for this measure and 'n' signifies participants evaluable for specified category.
Measure: Number; unit: participants
Arm/Group | Etanercept
Number analyzed (Participants) | 4842
participants
  AEs: Without Concomitant MTX (n = 2387) | 1145
  SAEs: Without Concomitant MTX (n = 2387) | 343
  AEs: With Concomitant MTX (n = 2455) | 1103
  SAEs: With Concomitant MTX (n = 2455) | 305

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 649/4871
Other Adverse Events (participants affected / at risk) | 1921/4871
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=4871)
Anaemia (Blood and lymphatic system disorders) | 7
Bone marrow failure (Blood and lymphatic system disorders) | 1
Bone marrow toxicity (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 4
Lymphadenitis (Blood and lymphatic system disorders) | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 2
Sideroblastic anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 6
Angina pectoris (Cardiac disorders) | 3
Aortic valve incompetence (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 18
Atrioventricular block second degree (Cardiac disorders) | 1
Bradyarrhythmia (Cardiac disorders) | 1
Bundle branch block right (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 11
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 7
Coronary artery stenosis (Cardiac disorders) | 2
Coronary artery thrombosis (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Intracardiac thrombus (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 4
Myocardial infarction (Cardiac disorders) | 7
Myocarditis (Cardiac disorders) | 1
Myocarditis post infection (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pulmonary valve incompetence (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 5
Tachycardia (Cardiac disorders) | 2
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Spondylolisthesis (Congenital, familial and genetic disorders) | 1
Von Willebrand's disease (Congenital, familial and genetic disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Vestibular neuronitis (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 2
Hyperparathyroidism secondary (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Toxic nodular goitre (Endocrine disorders) | 1
Cataract (Eye disorders) | 2
Chorioretinopathy (Eye disorders) | 1
Dacryoadenitis acquired (Eye disorders) | 1
Keratoconjunctivitis sicca (Eye disorders) | 1
Macular degeneration (Eye disorders) | 1
Optic ischaemic neuropathy (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Visual disturbance (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Appendicitis perforated (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 3
Colitis ulcerative (Gastrointestinal disorders) | 2
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Diverticular perforation (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 4
Leukoplakia oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Pancreatitis (Gastrointestinal disorders) | 3
Pancreatitis chronic (Gastrointestinal disorders) | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 3
Proctitis ulcerative (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 4
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 4
Chills (General disorders) | 2
Concomitant disease progression (General disorders) | 2
Condition aggravated (General disorders) | 76
Death (General disorders) | 3
Disease progression (General disorders) | 3
Drug effect decreased (General disorders) | 3
Drug ineffective (General disorders) | 14
Fatigue (General disorders) | 4
Gait disturbance (General disorders) | 2
General physical health deterioration (General disorders) | 6
Generalised oedema (General disorders) | 1
Impaired healing (General disorders) | 9
Inflammation of wound (General disorders) | 1
Injection site erythema (General disorders) | 1
Malaise (General disorders) | 1
Mass (General disorders) | 2
Multi-organ failure (General disorders) | 5
Necrosis (General disorders) | 1
Nodule (General disorders) | 1
Oedema mucosal (General disorders) | 1
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 5
Pyrexia (General disorders) | 6
Sudden cardiac death (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 2
Hepatomegaly (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 2
Abscess (Infections and infestations) | 4
Abscess intestinal (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Acid fast bacilli infection (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 4
Arthritis bacterial (Infections and infestations) | 2
Arthritis infective (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Body tinea (Infections and infestations) | 1
Breast abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Bronchopneumonia (Infections and infestations) | 3
Bursitis infective (Infections and infestations) | 2
Candida pneumonia (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Chlamydial infection (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Diabetic gangrene (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 5
Ear infection (Infections and infestations) | 1
Empyema (Infections and infestations) | 2
Endocarditis staphylococcal (Infections and infestations) | 2
Enterocolitis bacterial (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 3
Escherichia infection (Infections and infestations) | 4
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 5
Gastroenteritis Norwalk virus (Infections and infestations) | 1
Gastroenteritis rotavirus (Infections and infestations) | 2
Gastrointestinal infection (Infections and infestations) | 1
Genital abscess (Infections and infestations) | 1
Helicobacter gastritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 9
Herpes zoster ophthalmic (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Infected cyst (Infections and infestations) | 1
Infection (Infections and infestations) | 4
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 2
Klebsiella infection (Infections and infestations) | 2
Liver abscess (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Meningitis staphylococcal (Infections and infestations) | 1
Myringitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Necrotising fasciitis (Infections and infestations) | 1
Neuroborreliosis (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 3
Otitis media (Infections and infestations) | 2
Phlebitis infective (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 2
Pleural infection bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 24
Pneumonia bacterial (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 3
Pyoderma (Infections and infestations) | 2
Pyothorax (Infections and infestations) | 2
Relapsing fever (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 7
Septic arthritis staphylococcal (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 4
Staphylococcal sepsis (Infections and infestations) | 3
Stenotrophomonas infection (Infections and infestations) | 2
Streptococcal infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 2
Superinfection (Infections and infestations) | 1
Superinfection bacterial (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 8
Urosepsis (Infections and infestations) | 7
Vulval abscess (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 5
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 6
Device dislocation (Injury, poisoning and procedural complications) | 1
Device failure (Injury, poisoning and procedural complications) | 1
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1
Failure of implant (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 27
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 5
Forearm fracture (Injury, poisoning and procedural complications) | 2
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 3
Head injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2
Incision site erythema (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 2
Ligament rupture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 3
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 7
Meniscus lesion (Injury, poisoning and procedural complications) | 3
Muscle rupture (Injury, poisoning and procedural complications) | 1
Optic nerve injury (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 4
Post procedural complication (Injury, poisoning and procedural complications) | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Pubic rami fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 1
Synovial rupture (Injury, poisoning and procedural complications) | 2
Tendon rupture (Injury, poisoning and procedural complications) | 5
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2
Tibia fracture (Injury, poisoning and procedural complications) | 5
Upper limb fracture (Injury, poisoning and procedural complications) | 4
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood pressure abnormal (Investigations) | 1
Blood pressure increased (Investigations) | 2
Hepatic enzyme increased (Investigations) | 4
Transaminases increased (Investigations) | 2
Urine analysis abnormal (Investigations) | 1
Weight decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2
Diabetic foot (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Lactose intolerance (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 9
Cartilage development disorder (Musculoskeletal and connective tissue disorders) | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 5
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 16
Joint destruction (Musculoskeletal and connective tissue disorders) | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 5
Juvenile arthritis (Musculoskeletal and connective tissue disorders) | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 21
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 6
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Polyarthritis (Musculoskeletal and connective tissue disorders) | 4
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 75
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2
Spinal disorder (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 9
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 2
Cerebral ventricle dilatation (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 7
Cerebrovascular disorder (Nervous system disorders) | 1
Complex regional pain syndrome (Nervous system disorders) | 2
Critical illness polyneuropathy (Nervous system disorders) | 1
Cubital tunnel syndrome (Nervous system disorders) | 1
Demyelination (Nervous system disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysaesthesia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Essential tremor (Nervous system disorders) | 1
Facial paresis (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 2
Intercostal neuralgia (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Nerve compression (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Paresis (Nervous system disorders) | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 2
Quadriparesis (Nervous system disorders) | 1
Radicular pain (Nervous system disorders) | 1
Radicular syndrome (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 3
Ruptured cerebral aneurysm (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 4
Tarsal tunnel syndrome (Nervous system disorders) | 1
Thalamic infarction (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 1
Vascular encephalopathy (Nervous system disorders) | 1
Vasculitis cerebral (Nervous system disorders) | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1
Adjustment disorder (Psychiatric disorders) | 1
Alcohol abuse (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Restlessness (Psychiatric disorders) | 3
Schizophrenia (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 2
Acute prerenal failure (Renal and urinary disorders) | 5
Calculus bladder (Renal and urinary disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Crush syndrome (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Nephropathy toxic (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 4
Renal failure acute (Renal and urinary disorders) | 6
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Uterine disorder (Reproductive system and breast disorders) | 1
Uterine malposition (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1
Cutis laxa (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 4
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Abdominal operation (Surgical and medical procedures) | 1
Ankle arthroplasty (Surgical and medical procedures) | 1
Arthrodesis (Surgical and medical procedures) | 6
Bunion operation (Surgical and medical procedures) | 3
Cardioversion (Surgical and medical procedures) | 1
Cataract operation (Surgical and medical procedures) | 1
Cholecystectomy (Surgical and medical procedures) | 2
Ciliary body operation (Surgical and medical procedures) | 1
Colostomy closure (Surgical and medical procedures) | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1
Elbow operation (Surgical and medical procedures) | 1
Eye operation (Surgical and medical procedures) | 2
Foot operation (Surgical and medical procedures) | 4
Gastric bypass (Surgical and medical procedures) | 1
Hip arthroplasty (Surgical and medical procedures) | 6
Hysterectomy (Surgical and medical procedures) | 2
Intervertebral disc operation (Surgical and medical procedures) | 1
Joint arthroplasty (Surgical and medical procedures) | 3
Knee arthroplasty (Surgical and medical procedures) | 14
Retinopexy (Surgical and medical procedures) | 1
Skin graft (Surgical and medical procedures) | 1
Spinal corpectomy (Surgical and medical procedures) | 1
Spinal fusion surgery (Surgical and medical procedures) | 1
Spinal laminectomy (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 3
Stent placement (Surgical and medical procedures) | 1
Synovectomy (Surgical and medical procedures) | 8
Synoviorthesis (Surgical and medical procedures) | 2
Tendon operation (Surgical and medical procedures) | 1
Tendon sheath incision (Surgical and medical procedures) | 1
Toe operation (Surgical and medical procedures) | 2
Tonsillectomy (Surgical and medical procedures) | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1
Aneurysm (Vascular disorders) | 1
Aortic arteriosclerosis (Vascular disorders) | 1
Arterial disorder (Vascular disorders) | 1
Arterial thrombosis limb (Vascular disorders) | 1
Blood pressure inadequately controlled (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 8
Femoral arterial stenosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 5
Hypotension (Vascular disorders) | 1
Ischaemia (Vascular disorders) | 1
Pelvic venous thrombosis (Vascular disorders) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 7
Peripheral ischaemia (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 4
Vasculitis (Vascular disorders) | 2
Vasospasm (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 2
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=4871)
Anaemia (Blood and lymphatic system disorders) | 9
Eosinophilia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 8
Lymphadenopathy (Blood and lymphatic system disorders) | 6
Pancytopenia (Blood and lymphatic system disorders) | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Angina pectoris (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 5
Atrial fibrillation (Cardiac disorders) | 4
Cardiac discomfort (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 5
Cardiomegaly (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 6
Coronary artery insufficiency (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 14
Pericardial effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 6
Coarctation of the aorta (Congenital, familial and genetic disorders) | 1
Spondylolisthesis (Congenital, familial and genetic disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Ear haemorrhage (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Inner ear disorder (Ear and labyrinth disorders) | 1
Meniere's disease (Ear and labyrinth disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 6
Hyperthyroidism (Endocrine disorders) | 2
Toxic nodular goitre (Endocrine disorders) | 1
Abnormal sensation in eye (Eye disorders) | 2
Cataract (Eye disorders) | 8
Conjunctivitis (Eye disorders) | 3
Corneal infiltrates (Eye disorders) | 1
Dacryoadenitis acquired (Eye disorders) | 1
Dry eye (Eye disorders) | 3
Erythema of eyelid (Eye disorders) | 1
Eye disorder (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Eye inflammation (Eye disorders) | 5
Eye irritation (Eye disorders) | 2
Eye pruritus (Eye disorders) | 2
Eye swelling (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 5
Foreign body sensation in eyes (Eye disorders) | 1
Glaucoma (Eye disorders) | 2
Iritis (Eye disorders) | 2
Keratitis (Eye disorders) | 2
Lacrimation increased (Eye disorders) | 1
Macular degeneration (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Scleritis (Eye disorders) | 1
Scotoma (Eye disorders) | 1
Sicca syndrome (Eye disorders) | 3
Ulcerative keratitis (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 4
Visual disturbance (Eye disorders) | 7
Abdominal discomfort (Gastrointestinal disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 13
Abdominal tenderness (Gastrointestinal disorders) | 3
Abnormal faeces (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 5
Ascites (Gastrointestinal disorders) | 1
Bowel movement irregularity (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 1
Coeliac artery compression syndrome (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Dental caries (Gastrointestinal disorders) | 1
Dental discomfort (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 50
Diverticulum intestinal (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 5
Duodenitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 3
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 5
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 2
Gingival blister (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 6
Glossodynia (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 4
Hiatus hernia (Gastrointestinal disorders) | 1
Ileal ulcer (Gastrointestinal disorders) | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 82
Oedema mouth (Gastrointestinal disorders) | 1
Oesophageal pain (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 2
Oral disorder (Gastrointestinal disorders) | 1
Oral mucosal blistering (Gastrointestinal disorders) | 1
Oral mucosal erythema (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Paraesthesia oral (Gastrointestinal disorders) | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 5
Reflux oesophagitis (Gastrointestinal disorders) | 1
Saliva altered (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 2
Stomach granuloma (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 7
Tongue coated (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 22
Application site erythema (General disorders) | 1
Application site pruritus (General disorders) | 2
Asthenia (General disorders) | 8
Chest discomfort (General disorders) | 6
Chest pain (General disorders) | 6
Chills (General disorders) | 10
Condition aggravated (General disorders) | 93
Drug ineffective (General disorders) | 6
Face oedema (General disorders) | 3
Fat tissue increased (General disorders) | 1
Fatigue (General disorders) | 33
Feeling abnormal (General disorders) | 1
Feeling hot (General disorders) | 5
Gait disturbance (General disorders) | 2
General physical health deterioration (General disorders) | 6
Impaired healing (General disorders) | 4
Induration (General disorders) | 1
Inflammation (General disorders) | 2
Inflammation of wound (General disorders) | 1
Influenza like illness (General disorders) | 3
Injection site bruising (General disorders) | 1
Injection site erythema (General disorders) | 268
Injection site extravasation (General disorders) | 2
Injection site hypersensitivity (General disorders) | 16
Injection site induration (General disorders) | 10
Injection site inflammation (General disorders) | 2
Injection site irritation (General disorders) | 17
Injection site macule (General disorders) | 1
Injection site pain (General disorders) | 12
Injection site papule (General disorders) | 1
Injection site pruritus (General disorders) | 98
Injection site rash (General disorders) | 16
Injection site reaction (General disorders) | 69
Injection site swelling (General disorders) | 25
Injection site urticaria (General disorders) | 13
Injection site warmth (General disorders) | 6
Irritability (General disorders) | 2
Local reaction (General disorders) | 4
Local swelling (General disorders) | 3
Malaise (General disorders) | 7
Mucosal dryness (General disorders) | 4
Mucosal inflammation (General disorders) | 4
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 26
Pain (General disorders) | 13
Performance status decreased (General disorders) | 3
Prostration (General disorders) | 1
Pyrexia (General disorders) | 28
Rebound effect (General disorders) | 1
Sensation of foreign body (General disorders) | 3
Sense of oppression (General disorders) | 1
Swelling (General disorders) | 3
Tenderness (General disorders) | 2
Thirst (General disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 2
Hepatotoxicity (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 13
Abscess (Infections and infestations) | 1
Abscess jaw (Infections and infestations) | 4
Acute tonsillitis (Infections and infestations) | 7
Arthritis bacterial (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 1
Borrelia infection (Infections and infestations) | 3
Breast abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 107
Bronchitis bacterial (Infections and infestations) | 6
Bronchopneumonia (Infections and infestations) | 3
Campylobacter infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 2
Conjunctivitis bacterial (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Cystitis (Infections and infestations) | 20
Diverticulitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Ear infection bacterial (Infections and infestations) | 1
Eczema infected (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 7
Erythema infectiosum (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Eye infection bacterial (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 13
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 5
Fungal skin infection (Infections and infestations) | 5
Furuncle (Infections and infestations) | 8
Gastroenteritis (Infections and infestations) | 9
Gastroenteritis Norwalk virus (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 3
Gastrointestinal candidiasis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 19
Genital abscess (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Genital infection fungal (Infections and infestations) | 2
Gingival infection (Infections and infestations) | 2
Groin abscess (Infections and infestations) | 2
Helicobacter gastritis (Infections and infestations) | 3
Herpes ophthalmic (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 5
Herpes virus infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 22
Herpes zoster ophthalmic (Infections and infestations) | 1
Infected insect bite (Infections and infestations) | 1
Infection (Infections and infestations) | 27
Infection in an immunocompromised host (Infections and infestations) | 6
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Injection site cellulitis (Infections and infestations) | 1
Injection site pustule (Infections and infestations) | 3
Laryngitis (Infections and infestations) | 6
Lobar pneumonia (Infections and infestations) | 1
Localised infection (Infections and infestations) | 4
Lung infection (Infections and infestations) | 1
Lymph node abscess (Infections and infestations) | 1
Lymphangitis (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 163
Onychomycosis (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 4
Oral fungal infection (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 9
Oropharyngeal candidiasis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 2
Otitis media (Infections and infestations) | 5
Paronychia (Infections and infestations) | 5
Parotitis (Infections and infestations) | 1
Perianal fungal infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 6
Pharyngitis bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 17
Pneumonia haemophilus (Infections and infestations) | 1
Pulpitis dental (Infections and infestations) | 1
Pyelocystitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Pyoderma (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 11
Respiratory tract infection (Infections and infestations) | 45
Rhinitis (Infections and infestations) | 13
Scarlet fever (Infections and infestations) | 1
Sinobronchitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 37
Skin bacterial infection (Infections and infestations) | 2
Skin infection (Infections and infestations) | 3
Soft tissue infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 2
Subcutaneous abscess (Infections and infestations) | 4
Tinea pedis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 5
Tooth abscess (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 4
Tracheobronchitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 49
Upper respiratory tract infection bacterial (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 29
Urogenital trichomoniasis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Vaginal candidiasis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Viral infection (Infections and infestations) | 3
Viral upper respiratory tract infection (Infections and infestations) | 3
Vulvovaginal mycotic infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Accident at work (Injury, poisoning and procedural complications) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 3
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 20
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 6
Forearm fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2
Injury (Injury, poisoning and procedural complications) | 4
Joint dislocation (Injury, poisoning and procedural complications) | 4
Joint injury (Injury, poisoning and procedural complications) | 2
Joint sprain (Injury, poisoning and procedural complications) | 5
Ligament rupture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2
Open wound (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 3
Rib fracture (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 2
Seroma (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Skin injury (Injury, poisoning and procedural complications) | 4
Skin laceration (Injury, poisoning and procedural complications) | 2
Splinter (Injury, poisoning and procedural complications) | 1
Stress fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2
Thermal burn (Injury, poisoning and procedural complications) | 3
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Venomous sting (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 2
Wrist fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 13
Arthroscopy (Investigations) | 6
Aspartate aminotransferase increased (Investigations) | 2
Beta globulin increased (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood albumin increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 1
Blood creatine increased (Investigations) | 1
Blood creatinine increased (Investigations) | 9
Blood glucose increased (Investigations) | 4
Blood phosphorus decreased (Investigations) | 1
Blood pressure increased (Investigations) | 5
Blood smear test abnormal (Investigations) | 1
Blood urine present (Investigations) | 1
Body temperature increased (Investigations) | 5
C-reactive protein increased (Investigations) | 3
Cardiac murmur (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 9
Glycosylated haemoglobin increased (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Heart rate increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 2
Hysteroscopy (Investigations) | 1
Intraocular pressure increased (Investigations) | 1
Investigation (Investigations) | 1
Laparoscopy (Investigations) | 1
Liver function test abnormal (Investigations) | 19
Low density lipoprotein increased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Mean cell volume increased (Investigations) | 2
Monocyte count increased (Investigations) | 2
Mycobacteria blood test positive (Investigations) | 1
N-terminal pro-brain natriuretic peptide (NT-proBNP) (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Nitrite urine present (Investigations) | 1
Platelet count decreased (Investigations) | 3
Protein total increased (Investigations) | 1
Red blood cell count decreased (Investigations) | 2
Red blood cell sedimentation rate increased (Investigations) | 2
Red cell distribution width increased (Investigations) | 1
Streptococcal identification test positive (Investigations) | 1
Thyroid gland scan abnormal (Investigations) | 1
Transaminases increased (Investigations) | 25
Tuberculosis test positive (Investigations) | 2
Vitamin C increased (Investigations) | 1
Vitamin D decreased (Investigations) | 1
Weight decreased (Investigations) | 5
Weight increased (Investigations) | 14
White blood cell count (Investigations) | 1
White blood cell count increased (Investigations) | 5
White blood cells urine positive (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Fluid retention (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 3
Xanthelasma (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 27
Arthritis (Musculoskeletal and connective tissue disorders) | 7
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 24
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 11
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 2
Dactylitis (Musculoskeletal and connective tissue disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Foot deformity (Musculoskeletal and connective tissue disorders) | 10
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 13
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 10
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 8
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 20
Kyphosis (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Lordosis (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 16
Myosclerosis (Musculoskeletal and connective tissue disorders) | 3
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 20
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 44
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 15
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2
Scleroderma (Musculoskeletal and connective tissue disorders) | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Synovial cyst (Musculoskeletal and connective tissue disorders) | 5
Synovitis (Musculoskeletal and connective tissue disorders) | 5
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 3
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 2
Benign neoplasm of cervix uteri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lentigo (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Ageusia (Nervous system disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Burning sensation (Nervous system disorders) | 7
Carotid arteriosclerosis (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 2
Cervical root pain (Nervous system disorders) | 2
Cervicobrachial syndrome (Nervous system disorders) | 1
Cervicogenic headache (Nervous system disorders) | 1
Cluster headache (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 54
Dizziness postural (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 49
Hemicephalalgia (Nervous system disorders) | 1
Hyperaesthesia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 16
Intercostal neuralgia (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 3
Mental impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Nerve root compression (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 20
Parosmia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Radial nerve palsy (Nervous system disorders) | 1
Reduced dexterity (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 8
Sensory disturbance (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Syncope vasovagal (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Vascular encephalopathy (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 7
Agitation (Psychiatric disorders) | 6
Alcohol abuse (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 5
Anxiety disorder (Psychiatric disorders) | 1
Aversion (Psychiatric disorders) | 2
Depressed mood (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 12
Hallucination (Psychiatric disorders) | 1
Initial insomnia (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Middle insomnia (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 2
Panic attack (Psychiatric disorders) | 2
Psychogenic pain disorder (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 8
Stress (Psychiatric disorders) | 1
Acute prerenal failure (Renal and urinary disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 3
Haematuria (Renal and urinary disorders) | 2
IgA nephropathy (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 3
Nephritis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Renal failure chronic (Renal and urinary disorders) | 2
Urge incontinence (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2
Erectile dysfunction (Reproductive system and breast disorders) | 2
Genital erythema (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Menstrual disorder (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Orchitis noninfective (Reproductive system and breast disorders) | 1
Ovarian adhesion (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 2
Prostatitis (Reproductive system and breast disorders) | 1
Pruritus genital (Reproductive system and breast disorders) | 1
Uterine cyst (Reproductive system and breast disorders) | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal erythema (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 6
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 28
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 1
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 2
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Pleural rub (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 6
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 31
Alopecia areata (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 6
Blood blister (Skin and subcutaneous tissue disorders) | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 25
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 3
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 10
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 6
Eczema weeping (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 68
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Female pattern baldness (Skin and subcutaneous tissue disorders) | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 19
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1
Melanosis (Skin and subcutaneous tissue disorders) | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 76
Pruritus allergic (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 15
Psoriasis (Skin and subcutaneous tissue disorders) | 11
Purpura (Skin and subcutaneous tissue disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 47
Rash erythematous (Skin and subcutaneous tissue disorders) | 3
Rash generalised (Skin and subcutaneous tissue disorders) | 10
Rash macular (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Rash papular (Skin and subcutaneous tissue disorders) | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 10
Rash vesicular (Skin and subcutaneous tissue disorders) | 2
Rosacea (Skin and subcutaneous tissue disorders) | 1
Scar (Skin and subcutaneous tissue disorders) | 1
Scar pain (Skin and subcutaneous tissue disorders) | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 2
Skin burning sensation (Skin and subcutaneous tissue disorders) | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 5
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 2
Skin inflammation (Skin and subcutaneous tissue disorders) | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 3
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 16
Skin swelling (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 15
Skin warm (Skin and subcutaneous tissue disorders) | 3
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 7
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 15
Ankle operation (Surgical and medical procedures) | 1
Apicectomy (Surgical and medical procedures) | 1
Arthrectomy (Surgical and medical procedures) | 1
Arthrodesis (Surgical and medical procedures) | 9
Bladder neoplasm surgery (Surgical and medical procedures) | 1
Bone lesion excision (Surgical and medical procedures) | 1
Bunion operation (Surgical and medical procedures) | 4
Bursa removal (Surgical and medical procedures) | 1
Cataract operation (Surgical and medical procedures) | 4
Catheterisation cardiac (Surgical and medical procedures) | 1
Colostomy closure (Surgical and medical procedures) | 1
Corneal transplant (Surgical and medical procedures) | 1
Dental implantation (Surgical and medical procedures) | 2
Dental operation (Surgical and medical procedures) | 9
Dental treatment (Surgical and medical procedures) | 2
Endodontic procedure (Surgical and medical procedures) | 1
Eye operation (Surgical and medical procedures) | 1
Fasciectomy (Surgical and medical procedures) | 1
Female sterilisation (Surgical and medical procedures) | 1
Foot operation (Surgical and medical procedures) | 11
Hip arthroplasty (Surgical and medical procedures) | 14
Hip surgery (Surgical and medical procedures) | 1
Hospitalisation (Surgical and medical procedures) | 21
Hysterectomy (Surgical and medical procedures) | 2
Inguinal hernia repair (Surgical and medical procedures) | 1
Joint arthroplasty (Surgical and medical procedures) | 2
Knee arthroplasty (Surgical and medical procedures) | 10
Knee operation (Surgical and medical procedures) | 1
Limb operation (Surgical and medical procedures) | 1
Malignant tumour excision (Surgical and medical procedures) | 1
Meniscus removal (Surgical and medical procedures) | 1
Myomectomy (Surgical and medical procedures) | 1
Nail operation (Surgical and medical procedures) | 1
Nasal cyst removal (Surgical and medical procedures) | 1
Nasal operation (Surgical and medical procedures) | 1
Osteotomy (Surgical and medical procedures) | 2
Palatal operation (Surgical and medical procedures) | 1
Peripheral nerve destruction (Surgical and medical procedures) | 1
Prostatectomy (Surgical and medical procedures) | 1
Rehabilitation therapy (Surgical and medical procedures) | 2
Removal of internal fixation (Surgical and medical procedures) | 4
Renal stone removal (Surgical and medical procedures) | 1
Rheumatoid nodule removal (Surgical and medical procedures) | 1
Shoulder arthroplasty (Surgical and medical procedures) | 4
Sinus operation (Surgical and medical procedures) | 1
Skin neoplasm excision (Surgical and medical procedures) | 1
Spinal decompression (Surgical and medical procedures) | 1
Spinal laminectomy (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 3
Synovectomy (Surgical and medical procedures) | 23
Synoviorthesis (Surgical and medical procedures) | 3
Tendon operation (Surgical and medical procedures) | 1
Tendon sheath incision (Surgical and medical procedures) | 3
Tendon sheath lesion excision (Surgical and medical procedures) | 3
Therapeutic procedure (Surgical and medical procedures) | 2
Toe operation (Surgical and medical procedures) | 2
Tooth extraction (Surgical and medical procedures) | 5
Uterine dilation and curettage (Surgical and medical procedures) | 1
Varicose vein operation (Surgical and medical procedures) | 1
Vascular stent insertion (Surgical and medical procedures) | 1
Wisdom teeth removal (Surgical and medical procedures) | 3
Wrist surgery (Surgical and medical procedures) | 1
Blood pressure fluctuation (Vascular disorders) | 2
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Flushing (Vascular disorders) | 4
Haematoma (Vascular disorders) | 11
Hot flush (Vascular disorders) | 5
Hypertension (Vascular disorders) | 21
Hypertensive crisis (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 5
Pallor (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 4
Thrombosis (Vascular disorders) | 4
Varicose vein (Vascular disorders) | 8
Vasculitis (Vascular disorders) | 2
Venous thrombosis (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Prioritization of endpoints as primary or secondary was not specified in protocol and was based on study team's inputs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.